CLINICAL TRIAL: NCT02893163
Title: CHANGE (Canadian Health Advanced by Nutrition and Graded Exercise) Cancer Alberta: A Primary Care Program for Cancer Prevention and Screening
Brief Title: CHANGE Cancer Alberta: A Primary Care Program for Cancer Prevention and Screening
Acronym: CHANGECaAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Alberta Innovates Health Solutions (Other); Alberta Pulse Growers (Other); Alberta Health services (Other); Metabolic Syndrome Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00058125
Record Dates: First submitted 2016-08-22; First posted 2016-09-08 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Metabolic Syndrome; Risk Factors
Keywords: Metabolic Syndrome; Cancer Risk; Lifestyle Interventions; Primary Care; Behavioural Change
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHANGE Intervention (Experimental): The CHANGE intervention is a personalized approach to nutrition and exercise modification supported by a interdisciplinary team. The FD will recruit patients, complete baseline measurements and stabilize medication. The RD will create a diet plan tailored to the individual patient based on the intervention protocol. The ES will create an exercise plan tailored to the individual patient based on the intervention protocol. At the start, patients will meet weekly with the RD and ES in order to monitor progress, ascertain barriers and facilitators to change, and ensure adherence for the first 12 weeks of the intervention. Meetings will then occur monthly for the remaining 9 months of the intervention. Visits with the FD will occur every 3 months for the 12 month intervention to monitor progress, encourage behaviour change. A follow-up visit with the Research Coordinator will take place at 18 months.
  Interventions: Behavioral: CHANGE Intervention
- Usual Care (Active Comparator): The usual care arm of the study will involve regular care from the patients' FD. This may involve discussions regarding nutrition and exercise. The FD will still recruit patients, complete baseline measurements and stabilize medication. Visits to the FD will occur as usual care dictates. Participating PCNs randomized to usual care will still have interdisciplinary team members available but the referral arrangements are and will continue to be ad hoc. For the study, we will mandate that control patients have follow-up with the Research Coordinator at 3, 12 and 18 months for the purpose of assessing outcomes. At these time points, appointments will not be scheduled with the FD to manage their disease; rather, the purpose of the visit is to just conduct the outcome assessment.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: CHANGE Intervention — Canadian Health Advanced by Nutrition and Graded Exercise Protocol
  Arms: CHANGE Intervention
Other: Usual Care — Usual Care by Family Doctor
  Arms: Usual Care

SUMMARY:
The primary purpose of this trial will be to test the effectiveness of CHANGE intervention to increase physical activity, improve diets, reduce obesity and reverse Metabolic Syndrome among adult patients identified as at risk for cancer due to diet and physical activity behaviours when implemented in typical primary care settings within the Alberta context.

DETAILED DESCRIPTION:
The study is a cluster randomized control trial of 16 Primary Care Networks (PCN) in Alberta. Inclusion and exclusion criteria will occur at both the cluster and the patient levels. Site criteria have been designed to ensure implementation of the intervention is possible while contamination to the control sites is minimized. Patient level criteria are designed to include as many patients with Metabolic Syndrome identified at risk for cancer due to diet and physical activity behaviours as possible, maximizing generalizability, while ensuring that patients recruited are safely able to follow the CHANGE intervention.

CHANGE intervention utilizes a novel approach of embedding the expertise of Dietitians (RD) and Exercise Specialists (ES) with a patient's own Family Doctor (FD) to support a personalized nutrition and exercise intervention for patients with Metabolic Syndrome identified at risk for cancer due to diet and physical activity behaviours that is feasible to implement across diverse practice settings. There is sufficient data to support that the individual components of lifestyle interventions (diet and exercise) are efficacious. Unfortunately, primary care currently has limited capacity to implement lifestyle interventions to manage individuals who are overweight or obese. Family Doctors experience various barriers to providing diet and exercise counseling, including lack of staff and resources, limited time for effective health promotion counseling and limited specialized training. In order to provide quality of care for patients with Metabolic Syndrome identified at risk for cancer due to diet and physical activity behaviours, the investigators need to reduce these barriers and support Family Doctors with health care professionals who have the skills and time to help patients change their behaviours.

Although access to interdisciplinary teams has increased in Alberta over the past few years through the development of Primary Care Networks, the optimal composition of these teams has not yet been determined. There is significant evidence to support increased diet and exercise professionals within these primary care teams. Currently, Primary Care Networks are making decisions on how to structure the health care team for their networks. This recent development and strong provincial organizational structure creates a unique time and location to conduct a trial examining the prevention activities of health care teams. Findings from the CHANGE Cancer Alberta Study will inform Primary Care Network business plans to support the implementation of the CHANGE intervention broadly across Alberta.

ELIGIBILITY:
Inclusion Criteria:

Cluster level: Inclusion criteria: These include: 1) PCN within Alberta, 2) ability to incorporate RDs and ESs into the health care team.

Patient level: Inclusion criteria:

1. Adult patients (18+);
2. Adjusted BMI 26-40. This is a BMI calculated with the measured body weight minus 5 kg to reflect potential shifts in fluid balance;
3. Edmonton Obesity Stage 1 or 2(62). • Stage 1 patients have obesity-related subclinical risk factor(s) (e.g., borderline hypertension, impaired fasting glucose, elevated liver enzymes, Etc.), mild physical symptoms (e.g., dyspnea on moderate exertion, occasional aches and pains, fatigue, etc.), mild psychopathology, mild functional limitations and/or mild impairment of well being.

   • Stage 2 patients have established obesity-related chronic disease(s) (e.g., hypertension, type 2 diabetes, sleep apnea, osteoarthritis, reflux disease, polycystic ovary syndrome, anxiety disorder, etc.), moderate limitations in activities of daily living and/or well being.
4. Have Metabolic Syndrome (MetS is defined as having 3 of the 5 following criteria):

   1. Fasting Blood Glucose > 5.6 mmol/L or receiving pharmacotherapy;
   2. Blood Pressure of > 130/85 mm Hg or receiving pharmacotherapy;
   3. Triglyceride of > 1.7 mmol/L or receiving pharmacotherapy;
   4. HDL-C < 1.0 mmol/L Males and <1.3 mmol/L females;
   5. Increased Abdominal Circumference as per protocol.
5. Patients identified at risk for cancer due to diet and physical activity behaviours:

   a. Physical inactivity measured by: i. less than 150 minutes of moderate activity (i.e., brisk walking, bike riding, jogging) per week and/or strength trains less than 2 times weekly] OR ii. high sedentary time (>11 hours per day 1,2 ) AND b. Dietary behaviour risk measured by: i. Diabetes risk score of high or very high or fasting glucose or Hgb A1c above normal OR ii. Abnormal fasting plasma lipid profile AND c. 10-Year cardiovascular risk score >10%.

   -

Exclusion Criteria:

Cluster level: Exclusion criteria: Previous involvement of the CHANGE intervention.

Patient Level: Exclusion criteria: These include:

1. Edmonton Obesity Stage 0, 3, or 4(62).

   • Stage 0 patients have no apparent obesity-related risk factors, no physical symptoms, no psychopathology, no functional limitations and/or impairment of well being. They do not require intensive lifestyle interventions.

   • Stage 3 patients have established end-organ damage such as myocardial infarction, heart failure, diabetic complications, incapacitating osteoarthritis, significant psychopathology, significant functional limitation(s) and/or impairment of well being. This person requires intensive obesity treatment including pharmacological and surgical treatment options.

   • Stage 4 patients have severe (potentially end-stage) disability/ies from obesity-related chronic diseases, severe disabling psychopathology, severe functional limitation(s) and/or severe impairment of well being. Aggressive obesity management is required if feasible that includes palliative measures such as pain management, occupational therapy and psychosocial support.
2. Unable to speak, read or understand English.
3. Have a medical or physical condition that makes moderate intensity activity difficult or unsafe.
4. Diagnosis of Type 1 diabetes mellitus.
5. Type 2 diabetes only if any of the following are present

   o Proliferative diabetic retinopathy

   o Nephropathy (serum creatinine > 160 μmol/L)
   * Clinically manifest neuropathy defined as absent ankle jerks
   * Severe fasting hyperglycemia > 11 mmol/L
   * Peripheral vascular disease
6. Significant medical comorbidities, including uncontrolled metabolic disorders (e.g., thyroid, renal, liver), heart disease, stroke and ongoing substance abuse.
7. Clinically significant renal failure.
8. Diagnosis of cancer (other than non-melanoma skin cancer) that is currently being treated with radiation or chemotherapy.
9. Diagnosis of psychiatric disorders (cognitive impairment) that would limit adequate informed consent or ability to comply with study protocol.
10. Diagnosis of a terminal illness and/or in hospice care.
11. Pregnancy, lactating or planning to become pregnant during the study period.
12. Investigator discretion for clinical safety or protocol adherence reasons. This is based on the doctor's judgement. Patients whom the doctor believes will not be responsive to the intervention should be excluded.
13. Chronic inflammatory diseases. This includes clinically active inflammatory diseases such as clinically active ulcerative colitis, Crohn's disease or collagen vascular disease.
14. Patients currently attending an intensive lifestyle intervention (i.e. diabetes program, hypertension lipid clinic)

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2016-08; Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Primary Cancer Risk Outcome - Physical Activity | Baseline, 12 months
  Proportion of patients with improved physical activity levels (step counts) measured by 7-day accelerometer step count
Primary Cancer Risk Outcome - Nutrition | Baseline, 3 months. 12 months, 18 months
  Proportion of patients with improved eating behaviours (Healthy Eating Index) as measured by 2-24 hour dietary recalls
Primary Metabolic Syndrome Outcomes | Baseline, 3 months, 12 months, 18 months
  Proportion of patients achieving reversal of Metabolic Syndrome (no longer meeting 3 of 5 diagnostic criteria

SECONDARY OUTCOMES:
Secondary Cancer Risk Outcome - BMI | Baseline, 3 months, 12 months, 18 months
  Proportion of patients achieving reduction in BMI
Secondary Caner Risk Outcome - Waist Circumference | Baseline, 3 months, 12 months, 18 months
  Proportion of patients achieving reduction in waist circumference
Secondary Metabolic Syndrome Outcome - Cardiovascular Risk | Baseline, 3 months, 12 months, 18 months
  Proportion of patients achieving reduction in 10-year cardiovascular risk (as calculated by the PROCAM (Prospective Cardiovascular Munster Study) risk algorithm)

OTHER OUTCOMES:
Patient Self Reported Health | Baseline, 3 months, 12 months, 18 months
  Proportion of patients improving self-reported health (using the short-form-12 [SF-12 (Short Form-12) Health Scale Scoring]
Patient Self Reported Quality of Life | Baseline, 3 months, 12 months, 18 months
  Proportion of patients improving self-reported quality of life (using EQ-5D-5L (EuroQol-5 Dimension-5 Level))

CONTACTS AND LOCATIONS:
Overall Officials: Doug Klein, MD, MSc, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brauer P, Gorber SC, Shaw E, Singh H, Bell N, Shane ARE, Jaramillo A, Tonelli M; Canadian Task Force on Preventive Health Care. Recommendations for prevention of weight gain and use of behavioural and pharmacologic interventions to manage overweight and obesity in adults in primary care. CMAJ. 2015 Feb 17;187(3):184-195. doi: 10.1503/cmaj.140887. Epub 2015 Jan 26. No abstract available. PMID 25623643
- [Background] Petrella RJ, Lattanzio CN, Overend TJ. Physical activity counseling and prescription among canadian primary care physicians. Arch Intern Med. 2007 Sep 10;167(16):1774-81. doi: 10.1001/archinte.167.16.1774. PMID 17846397
- [Background] Petrella RJ, Koval JJ, Cunningham DA, Paterson DH. Can primary care doctors prescribe exercise to improve fitness? The Step Test Exercise Prescription (STEP) project. Am J Prev Med. 2003 May;24(4):316-22. doi: 10.1016/s0749-3797(03)00022-9. PMID 12726869
- [Background] Brown JB, Harris SB, Webster-Bogaert S, Wetmore S, Faulds C, Stewart M. The role of patient, physician and systemic factors in the management of type 2 diabetes mellitus. Fam Pract. 2002 Aug;19(4):344-9. doi: 10.1093/fampra/19.4.344. PMID 12110552
- [Background] Kirk SF, Tytus R, Tsuyuki RT, Sharma AM. Weight management experiences of overweight and obese Canadian adults: findings from a national survey. Chronic Dis Inj Can. 2012 Mar;32(2):63-9. PMID 22414302
- [Background] Dahrouge S, Dinh T. The economic impact of improvements in primary healthcare performance. [electronic resource]: Ottawa, Ont.] : Canadian Health Services Research Foundation, 2012 (Saint-Lazare, Quebec : Canadian Electronic Library, 2012); 2012.
- [Background] Tsai AG, Wadden TA. Treatment of obesity in primary care practice in the United States: a systematic review. J Gen Intern Med. 2009 Sep;24(9):1073-9. doi: 10.1007/s11606-009-1042-5. Epub 2009 Jun 27. PMID 19562419
- [Background] McAlister FA, Stewart S, Ferrua S, McMurray JJ. Multidisciplinary strategies for the management of heart failure patients at high risk for admission: a systematic review of randomized trials. J Am Coll Cardiol. 2004 Aug 18;44(4):810-9. doi: 10.1016/j.jacc.2004.05.055. PMID 15312864
- [Background] Singh S, Devanna S, Edakkanambeth Varayil J, Murad MH, Iyer PG. Physical activity is associated with reduced risk of esophageal cancer, particularly esophageal adenocarcinoma: a systematic review and meta-analysis. BMC Gastroenterol. 2014 May 30;14:101. doi: 10.1186/1471-230X-14-101. PMID 24886123
- [Background] Forman MR, Hursting SD, Umar A, Barrett JC. Nutrition and cancer prevention: a multidisciplinary perspective on human trials. Annu Rev Nutr. 2004;24:223-54. doi: 10.1146/annurev.nutr.24.012003.132315. PMID 15189120
- [Background] Perk J, De Backer G, Gohlke H, Graham I, Reiner Z, Verschuren M, Albus C, Benlian P, Boysen G, Cifkova R, Deaton C, Ebrahim S, Fisher M, Germano G, Hobbs R, Hoes A, Karadeniz S, Mezzani A, Prescott E, Ryden L, Scherer M, Syvanne M, Scholte op Reimer WJ, Vrints C, Wood D, Zamorano JL, Zannad F; European Association for Cardiovascular Prevention & Rehabilitation (EACPR); ESC Committee for Practice Guidelines (CPG). European Guidelines on cardiovascular disease prevention in clinical practice (version 2012). The Fifth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of nine societies and by invited experts). Eur Heart J. 2012 Jul;33(13):1635-701. doi: 10.1093/eurheartj/ehs092. Epub 2012 May 3. No abstract available. PMID 22555213
- [Background] Handelsman Y, Mechanick JI, Blonde L, Grunberger G, Bloomgarden ZT, Bray GA, Dagogo-Jack S, Davidson JA, Einhorn D, Ganda O, Garber AJ, Hirsch IB, Horton ES, Ismail-Beigi F, Jellinger PS, Jones KL, Jovanovic L, Lebovitz H, Levy P, Moghissi ES, Orzeck EA, Vinik AI, Wyne KL; AACE Task Force for Developing a Diabetes Comprehensive Care Plan. American Association of Clinical Endocrinologists Medical Guidelines for clinical practice for developing a diabetes mellitus comprehensive care plan: executive summary. Endocr Pract. 2011 Mar-Apr;17(2):287-302. doi: 10.4158/ep.17.2.287. No abstract available. PMID 21474421
- [Background] Brenner DR. Cancer incidence due to excess body weight and leisure-time physical inactivity in Canada: implications for prevention. Prev Med. 2014 Sep;66:131-9. doi: 10.1016/j.ypmed.2014.06.018. Epub 2014 Jun 23. PMID 24967956